CLINICAL TRIAL: NCT05793190
Title: Feal Mycobiome Profiling Depending on Alcoholic Liver Disease Severity.
Brief Title: Gut Mycobiome Profile in Alcoholic Liver Disease.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GMALD
Record Dates: First submitted 2023-03-19; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Alcoholic Liver Disease
MeSH Terms: conditions — Liver Diseases, Alcoholic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Mycobial DNA were isolated from collected fecal samples by using DNeasy powersoil pro kit and subjected for nuclear ribosomal RNA internal transcribed spacer (ITS) gene sequencing were performed using the MiSeq sequencer on the illumine platform
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Healthy Control: Total number of 20 Healthy Control participants Included in the study
- Alcoholic hepatitis: Total number of 30 Alcoholic hepatitis patients included in the study
- Alcoholic cirrhosis: Total number of 30 alcoholic cirrhosis patients included in the study
- Acute-on-Chronic Liver Failure: Total number of 15 alcoholic acute-on-chronic liver failure patients included in the study
- Alcoholic Hepatocellular carcinoma: Total number of 25 Alcoholic Hepatocellular carcinoma patients included in the study

SUMMARY:
The fecal mycobiome, which refers to the community of fungi that resides in the human gut, is an important component of the gut microbiome. Research has shown that changes in the gut microbiome, including alterations in the fecal mycobiome, may play a role in the development and progression of alcoholic liver disease (ALD).One study published in the journal Gut Microbes found that individuals with ALD had a different gut microbiome composition compared to healthy individuals, including alterations in the levels of certain fungal species. Specifically, the study found that there was an increase in the abundance of the fungal genus Saccharomyces in individuals with ALD. This is significant because Saccharomyces is known to produce ethanol, which can contribute to liver damage in individuals with ALD.Another study published in the journal PLOS One found that there were differences in the levels of fungal metabolites in the fecal samples of individuals with ALD compared to healthy individuals. Specifically, the study found that there were higher levels of certain fungal metabolites, including acetaldehyde and ethanol, in the fecal samples of individuals with ALD.These findings suggest that the fecal mycobiome may play an important role in the development and progression of ALD. Maintaining a healthy gut microbiome through a balanced diet and other lifestyle factors may be an important strategy for preventing and managing ALD, and further research into the role of the fecal mycobiome in this condition is warranted.

DETAILED DESCRIPTION:
Fecal samples were collected prospectively from 120 participants including Healthy Control (HC=20), Alcoholic hepatitis (AH=30), alcoholic cirrhosis (AC=30), Acute-on-Chronic Liver Failure (ACLF=15), Alcoholic Hepatocellular carcinoma (AHCC=25). Mycobial DNA were isolated from collected fecal samples by using DNeasy powersoil pro kit and subjected for nuclear ribosomal RNA internal transcribed spacer (ITS) gene sequencing were performed using the MiSeq sequencer on the illumine platform and based on the phylogenetic relationship, ITS-based Mycobiome Taxonomic Profiling was performed to discovery gut mycobial compositional shift along with ALD severity progression. To discover compositional shift along with ALD severity progression, various statistical analysis method is going to be performed which includes standard mean based differential analysis such ANOVA, Principle component analysis to established the basic compositional variation in all the groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to Chuncheon Sacred Hallym hospital with a diagnosis of ALD will be screened and potentially recruited.
* ALD patients will be identified based on the recent American Association of the Study of Liver Disease (AASLD) guidelines:

  1. onset of jaundice within 8 weeks,
  2. ongoing consumption of ethanol of >40 for women or >60 in men for 6 months or <60 days of abstinence before onset of jaundice,
  3. Aspartate transaminase (AST>50), AST:ALT>1.5 and both <400 IU/L,
  4. Total bilirubin >3, or liver biopsy showing histologic features of ALD.

Exclusion Criteria:

* If patients have a history of inflammatory bowel disease, irritable bowel syndrome, gastrointestinal malignancy, or gastrointestinal surgery.
* Patients with acute pancreatitis or history of chronic pancreatitis will also be excluded. The diagnosis of acute pancreatitis and chronic pancreatitis will be ascertained from their history and physical.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Total number of 500 participants were enrolled in this clinical trial, out those 500 participants only 120 were met with the inclusion criteria therefore 380 participants were excluded from this clicial trial. Fecal samples were collected prospectively from 120 participants including Healthy Control (HC=20), Alcoholic hepatitis (AH=30), alcoholic cirrhosis (AC=30), Acute-on-Chronic Liver Failure (ACLF=15), Alcoholic cirrhosis (AC=25).
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Gut mycobiome compositional signature in Alcoholic liver diseases | 2 years
  Research has shown that the gut mycobiome, which refers to the community of fungi that resides in the human gut, may have a distinct compositional signature in individuals with alcoholic liver disease (ALD). Microorganisms found that individuals with ALD had a higher abundance of certain fungal species, including Candida, Malassezia, and Saccharomyces, compared to healthy individuals and genus Saccharomyces. Saccharomyces is of particular interest in ALD as it is known to produce ethanol, which can contribute to liver damage in individuals with ALD. Furthermore, higher levels of certain fungal metabolites, including acetaldehyde and ethanol, in the fecal samples of individuals with ALD. These findings suggest that the gut mycobiome may play a role in the development and progression of ALD, and that alterations in the composition of the gut mycobiome may be a potential biomarker for this condition.
Gut mycobiome biomarkers identification for early detection of decompensated alcoholic liver disease | 2 years
  While there is still much research to be done, studies have identified potential gut mycobiome biomarkers that may be used for the early detection of ALD and its progression to more severe stages. Overall, previous findings suggest that the gut mycobiome may be a valuable source of biomarkers for the early detection of ALD. However, further research is needed to confirm the accuracy and reliability of these potential biomarkers and to determine the best approach for their clinical use.
Health beneficial Gut Mycobiome identification in alcoholic liver disease | 2 years
  While research has primarily focused on the detrimental effects of altered gut mycobiome composition in individuals with alcoholic liver disease (ALD), there is also evidence to suggest that certain fungal species may have health benefits and could potentially play a role in the prevention or treatment of ALD. The fungal genus Debaryomyces was present at higher levels in the fecal samples of healthy individuals compared to individuals with ALD. Fungal species Rhodotorula mucilaginosa was able to reduce liver damage in rats with ALD. Rhodotorula mucilaginosa and Debaryomyces has also been shown to have anti-inflammatory and antioxidant properties, which may contribute to its protective effects on the liver. These findings suggest that certain fungal species may have health benefits and could potentially be used in the prevention or treatment of ALD.

CONTACTS AND LOCATIONS:
Overall Officials: Ki Tae Suk, PhD, Principal Investigator — Chuncheon Sacred Hallym hospital
Locations (1):
- Department of Internal Medicine, Hallym University Chuncheon Sacred Heart Hospital, Chuncheon, Gangwondo, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Demir M, Lang S, Hartmann P, Duan Y, Martin A, Miyamoto Y, Bondareva M, Zhang X, Wang Y, Kasper P, Bang C, Roderburg C, Tacke F, Steffen HM, Goeser T, Kruglov A, Eckmann L, Starkel P, Fouts DE, Schnabl B. The fecal mycobiome in non-alcoholic fatty liver disease. J Hepatol. 2022 Apr;76(4):788-799. doi: 10.1016/j.jhep.2021.11.029. Epub 2021 Dec 10. PMID 34896404
- [Background] Hindson J. Distinct faecal mycobiome in patients with NAFLD. Nat Rev Gastroenterol Hepatol. 2022 Feb;19(2):79. doi: 10.1038/s41575-022-00576-z. No abstract available. PMID 35017674
- [Background] Mbaye B, Borentain P, Magdy Wasfy R, Alou MT, Armstrong N, Mottola G, Meddeb L, Ranque S, Gerolami R, Million M, Raoult D. Endogenous Ethanol and Triglyceride Production by Gut Pichia kudriavzevii, Candida albicans and Candida glabrata Yeasts in Non-Alcoholic Steatohepatitis. Cells. 2022 Oct 27;11(21):3390. doi: 10.3390/cells11213390. PMID 36359786
- [Background] Lang S, Duan Y, Liu J, Torralba MG, Kuelbs C, Ventura-Cots M, Abraldes JG, Bosques-Padilla F, Verna EC, Brown RS Jr, Vargas V, Altamirano J, Caballeria J, Shawcross D, Lucey MR, Louvet A, Mathurin P, Garcia-Tsao G, Ho SB, Tu XM, Bataller R, Starkel P, Fouts DE, Schnabl B. Intestinal Fungal Dysbiosis and Systemic Immune Response to Fungi in Patients With Alcoholic Hepatitis. Hepatology. 2020 Feb;71(2):522-538. doi: 10.1002/hep.30832. Epub 2019 Aug 20. PMID 31228214
- [Background] Zeng S, Schnabl B. Roles for the mycobiome in liver disease. Liver Int. 2022 Apr;42(4):729-741. doi: 10.1111/liv.15160. Epub 2022 Jan 17. PMID 34995410